CLINICAL TRIAL: NCT04117529
Title: Phenotypic and Functional Characterisation of Human B-cell Response in Pemphigus and Application to Other Auto-immune Diseases
Brief Title: Phenotypic and Functional Characterisation of Human B-cell Response in Pemphigus
Acronym: CaReLyBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP190199; 2019-A00533-54 (Other: ANSM - IDRCB number)
Record Dates: First submitted 2019-09-26; First posted 2019-10-07 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Pemphigus Vulgaris; Pemphigus Foliaceus
Keywords: Pemphigus Vulgaris; Pemphigus Foliaceus; B-cell; Dermatology
MeSH Terms: conditions — Pemphigus | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Pemphigus or other autoimmune diseases.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Collection of 2 blood sample : The first one at the inclusion in the study, the second one between 6 months and 9 months after the inclusion. The sample consists of 2 tubes of EthyleneDiamineTetraAcetic (EDTA) of 7 mL.

SUMMARY:
Pemphigus is a rare autoimmune disease involving skin and mucous membranes characterized by the production of pathogenic autoantibodies directed against desmosomal transmembrane glycoproteins belonging to the cadherin family,responsible for the disruption of desmosomes leading to the acantholysis phenomenon.Two main classical subtypes of pemphigus have been individualized:pemphigus vulgaris and foliaceus,in which pathogenic autoantibodies are directed against desmoglein 3 and 1 respectively.The knowledge about B-cell populations responsible for pemphigus activity increased a lot.In pemphigus patients,B-cell population was shown to comprise auto-reactive B lymphocytes producing antibodies targeting desmogleins,directly responsible for disease activity,and regulatory B lymphocytes.After rituximab treatment,clinical activity was proved to be associated with circulating auto-antibodies high titers and an increase of auto-reactive B-cells,whereas clinical remission was associated with a change in B-cell populations,as B cell repertoire changed from oligoclonal to polyclonal when reconstituting after treatment,with an increase of immatures and transitional B-cells producing IL-10.The mechanisms leading to autoreactive B-cells appearance,the precise role of B-reg in immune tolerance and the factors triggering the imbalance between pro autoimmune and regulatory immune B-cells leading to pemphigus activity remain to be discovered.Polymorphonuclear neutrophil granulocytes(PMN) are the first responders of the immune system to threats by invading microorganisms.Since 2004, PMN were shown to produce neutrophil extracellular traps(NET),structures consisting of decondensed chromatin embedded with histones,granular and cytoplasmic proteins that trap and kill microbes.In lupus recent works demonstrated evidences that NETs components are found in immune complexes responsible for tissue inflammation and that polyclonal activation of B-cell as well as memory B-cell activation could be obtain in presence of immune complexes derived from NET.Besides lupus,other works showed evidence of NETs implication in inflammatory and auto-immune states in rheumatoid arthritis and small vessel vasculitis.The hypotheses is that B-cell activation by NET might not be restricted to autoimmune diseases of which antibodies target NETs components.The aim is to assess the effects on B-cell activation and the phenotypic changes in B-cell population from pemphigus patients after stimulation by NET.

DETAILED DESCRIPTION:
Pemphigus is a rare autoimmune disease involving skin and mucous membranes with an incidence estimated as 0.7 to 7 new cases per million per year, responsible for non-negligible morbidity and mortality. Pemphigus is characterized by the production of pathogenic autoantibodies directed against two desmosomal proteins involved in keratinocyte adhesion (i.e. desmoglein 1 and desmoglein 3). These antibodies are responsible for the disruption of desmosomes leading to the acantholysis phenomenon, which results in the formation of skin and mucosal blisters. Two main classical subtypes of pemphigus have been individualized, pemphigus vulgaris (PV) and pemphigus foliaceus (PF), in which pathogenic autoantibodies are directed against desmosomal transmembrane glycoproteins belonging to the cadherin family, desmoglein 3, and desmoglein 1, respectively. As for many auto-immune diseases, high doses of corticosteroids (CS) remained the mainstay of first-line treatment for long time, alone or in conjunction with immunosuppressants. However, on these regimens, frequent relapses occurs when tapering CS dosage leading to long-term treatment and its associated risk of CS side effects.

Since ten years, the improvement in the knowledge of B-cell activation and survival, as well as their direct implication in auto-immune disease such as pemphigus through pathogenic auto-antibodies production, led to the identification of new therapeutic targets. New biological therapies based on B cell depletion were developed in severe autoimmune disorders, notably in pemphigus.

Several teams demonstrated the safety and efficacy of Rituximab, a chimeric immunoglobulin gamma-1(IgG1) monoclonal antibody(mAb) targeting the cluster of differentiation antigen 20(CD20) molecule expressed by normal B-cells from pre-B cells except for plasma cells, in severe pemphigus refractory to corticosteroids as well as in first line of treatment. Across these works, some of them concurred to improve the knowledge about B-cell populations responsible for pemphigus activity. In pemphigus patients, B-cell population was shown to comprise auto-reactive B lymphocytes producing antibodies targeting desmogleins, directly responsible for disease activity, and regulatory B lymphocytes (B-reg). After rituximab treatment of pemphigus patients, clinical activity was proved to be associated with circulating auto-antibodies high titers and an increase of auto-reactive B-cells, whereas clinical remission was associated with a change in B-cell populations, as B cell repertoire changed from oligoclonal to polyclonal when reconstituting after treatment, with an increase of immatures and transitional B-cells producing IL-10 (B-reg).

The mechanisms leading to autoreactive B-cells appearance, the precise role of B-reg in immune tolerance, and the factors triggering the imbalance between pro autoimmune and regulatory immune B-cells leading to pemphigus activity remain to be discovered. As for other auto-immune diseases, first flares and relapses were described following infectious events. Thus, infectious agents might trigger unknown mechanisms participating in the immune system imbalance by the activation of previously quiescent auto reactive B-cells or effector B-cells.

Polymorphonuclear neutrophil granulocytes (PMN) are the first responders of the immune system to threats by invading microorganisms; performing essential functions of innate immunity in host defence against a broad range of pathogens, notably by phagocytosis, intracellular degradation and extracellular discharge of antimicrobial factors. Since 2004, Polynuclear Neutral Neutrophil (PNN) were shown to produce neutrophil extracellular traps (NET), structures consisting of decondensed chromatin embedded with histones, granular and cytoplasmic proteins that trap and kill microbes. NET were initially consider to arise following cell death (NETosis) but NET formation was also described without PMN death with mitochondrial DNA extrusion. NET production during infectious events is responsible for the release of cytosolic, nuclear and mitochondrial antigens in the extracellular environment; this auto-antigen exposure constituting favourable conditions for autoimmune disease such as lupus erythematosus and AntiNeutrophil Cytoplasmic Antibody (ANCA) vasculitis, of which auto-antibodies targets belong to NET components (DNA, RNA, MPO, PR3). Besides antimicrobial function, an excessive production of NET or NET insufficient clearance were found to maintain tissue inflammation and excessive tissue damages that contribute to autoinflammatory and autoimmune diseases.

In lupus, recent works demonstrated evidences that NET components are found in immune complexes responsible for tissue inflammation and that polyclonal activation of B-cell as well as memory B-cell activation could be obtain in presence of immune complexes derived from NET.

Besides lupus, other works showed evidence of NET implication in inflammatory and auto-immune states in rheumatoid arthritis and small vessel vasculitis.

The investigators hypothesize that B-cell activation by NET might not be restricted to autoimmune diseases of which antibodies target NET components, as it is the case for lupus (DNA, RNA, LL37), Rheumatoid Arthritis(RA) (citrullinated proteins) or small vessel vasculitis (PR3, MPO).

Thus, the primary aim is to assess the effects on B-cell activation and the phenotypic changes in B-cell population from pemphigus patients after stimulation by neutrophil extracellular traps.

The secondary aim is to compare the results obtained in pemphigus patients to patients with other autoimmune diseases such as lupus, rheumatoid arthritis a Gougerot-Sjögren syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients man or woman
* Patients above 18 years old
* Patients fulfilling the diagnostic criteria for pemphigus (Lever et al, 1979), or for lupus (SLICC 2012), or for rheumatoid arthritis (ACR / EULAR 2009 criteria), or for Gougerot-Sjögren's syndrome (ACR criteria / EULAR 2016)
* Clinically active disease, defined by the presence of erosions or cutaneo-mucous bubbles for pemphigus, a SLEDAI score> 0 for lupus, a DAS28> 0 score for rheumatoid arthritis, and an EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score> 0 for Gougerot-Sjögren's syndrome
* Patients consenting to participate in the study
* Patients benefiting from the national healthcare insurance

Exclusion Criteria:

* Pregnant or lactating woman
* Patient already treated with biotherapy
* Patient already receiving treatment that may affect lymphocyte B populations: corticosteroid therapy> 10 mg / d or other immunosuppressant.
* Patient whose weight and / or hemoglobin level does not allow an additional blood sample during the assessment already provided by the treatment (according to the values in Appendix 2 of the Decree of April 12, 2018, which lists the research mentioned in 2 ° of Article L. 1121-1 of the Public Health Code)
* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Involvement of neutrophil extracellular traps (NETs) in the activation of B lymphocytes in Pemphigus | 9 months after inclusion
  This primary outcome measure is composite. It will be verified according to the following points : Measurement of activation parameters of total, auto-reactive, and regulator B lymphocytes of patients :
  * Quantification of membrane markers for activation of B lymphocytes (CD80, CD86, CD40)
  * Quantification of the production of pro-inflammatory cytokines (IL-6, IL-8, Tumor Necrosis Factor alpha (TNF alpha), IFNγ) by total and auto-reactive B lymphocytes
  * Quantification of the total production of immunoglobulins and antibodies specific for the disease
  * Quantification of IL-10 and Tumor Growth Factor (TGF) beta production by regulatory B cells.

SECONDARY OUTCOMES:
Demonstration that activation of the different sub-populations of B lymphocytes during NET exposure, if shown in pemphigus, is also in lupus, rheumatoid arthritis and Gougerot-Sjögren's syndrome relying on membrane markers for activation of B lymphocytes | 9 months after inclusion
  Quantification of membrane markers for activation of B lymphocytes (CD80, Cluster of Differentiation antigen 86 (CD86), CD40);
Demonstration that activation of the different sub-populations of B lymphocytes during NET exposure, if shown in pemphigus, is also lupus, rheumatoid arthritis and Gougerot-Sjögren's syndrome relying on pro-inflammatory cytokines | 9 months after inclusion
  Quantification of the production of pro-inflammatory cytokines (IL-6, IL-8, TNF-alpha(Tumor Necrosis Factor alpha), IFNγ) by total and auto-reactive B lymphocytes
Demonstration that activation of the different sub-populations of B lymphocytes during NET exposure, if shown in pemphigus, is also in lupus, rheumatoid arthritis and Gougerot-Sjögren's syndrome relying on immunoglobulins and antibodies | 9 months after inclusion
  Quantification of the total production of immunoglobulins and antibodies specific for the disease
Demonstration that activation of the different sub-populations of B lymphocytes during NET exposure, if shown in pemphigus,is also in lupus,rheumatoid arthritis and Gougerot-Sjögren's syndrome relying on IL-10 and TGFbeta production by regulatory B cells | 9 months after inclusion
  Quantification of IL-10 and TGFbeta production by regulatory B cells

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MUSETTE, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pr Philippe MUSETTE - Hôpital AVICENNE, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langan SM, Smeeth L, Hubbard R, Fleming KM, Smith CJ, West J. Bullous pemphigoid and pemphigus vulgaris--incidence and mortality in the UK: population based cohort study. BMJ. 2008 Jul 9;337(7662):a180. doi: 10.1136/bmj.a180. PMID 18614511
- [Background] Hashimoto T, Amagai M, Garrod DR, Nishikawa T. Immunofluorescence and immunoblot studies on the reactivity of pemphigus vulgaris and pemphigus foliaceus sera with desmoglein 3 and desmoglein 1. Epithelial Cell Biol. 1995;4(2):63-9. PMID 8688919
- [Background] Martel P, Joly P. Pemphigus: autoimmune diseases of keratinocyte's adhesion molecules. Clin Dermatol. 2001 Nov-Dec;19(6):662-74. doi: 10.1016/s0738-081x(00)00191-7. No abstract available. PMID 11705674
- [Background] Amagai M, Tsunoda K, Zillikens D, Nagai T, Nishikawa T. The clinical phenotype of pemphigus is defined by the anti-desmoglein autoantibody profile. J Am Acad Dermatol. 1999 Feb;40(2 Pt 1):167-70. doi: 10.1016/s0190-9622(99)70183-0. PMID 10025740
- [Background] Mahoney MG, Wang Z, Rothenberger K, Koch PJ, Amagai M, Stanley JR. Explanations for the clinical and microscopic localization of lesions in pemphigus foliaceus and vulgaris. J Clin Invest. 1999 Feb;103(4):461-8. doi: 10.1172/JCI5252. PMID 10021453